CLINICAL TRIAL: NCT02184585
Title: An Open-label, Randomized, Single Dose, Three-way Crossover Study to Determine the Bioavailability of Two Fixed Dose Combination Capsule Formulations of Dutasteride and Tamsulosin Hydrochloride (0.5mg/0.2mg) Relative to Co-administration of Dutasteride 0.5mg Capsules and Tamsulosin Hydrochloride 0.2mg Tablets in Healthy Male Subjects in the Fed and Fasted States
Brief Title: Comparative Bioavailability of Two Fixed Dose Combination (FDC) Formulations of Dutasteride and Tamsulosin Hydrochloride Relative to Co-administration of Dutasteride With Tamsulosin Hydrochloride in Healthy Male Subjects Under Fed and Fasted States
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 117057
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Prostatic Hyperplasia
Keywords: bioavailability; crossover design; healthy male volunteers; tamsulosin hydrochloride; Dutasteride
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1: Fasted state (Experimental): Treatment will be administered orally to 42 subjects in the fasted state. Subjects will be required to fast overnight (minimum 10 hours) and for a minimum of 4 hours after each dose. Subjects will participate in 3 treatment periods and assigned to one of six treatment sequences (ABC, ACB, BAC, BCA, CAB, CBA) in accordance with the randomization schedule generated by Clinical Statistics. The three treatment periods will be separated by a minimum washout period of 28 days
  Interventions: Drug: Treatment sequence A; Drug: Treatment sequence B; Drug: Treatment sequence C
- Cohort 2 : Fed state (Experimental): Treatment will be administered orally to 42 subjects in the fed state (high fat breakfast). Dosing will take place within 30 minutes of the start of the meal. Subjects will participate in 3 treatment periods and assigned to one of six treatment sequences (ABC, ACB, BAC, BCA, CAB, CBA) in accordance with the randomization schedule generated by Clinical Statistics. The three treatment periods will be separated by a minimum washout period of 28 days
  Interventions: Drug: Treatment sequence A; Drug: Treatment sequence B; Drug: Treatment sequence C

INTERVENTIONS:
Drug: Treatment sequence A — FDC 1 - Fixed dose combination capsule of dutasteride and tamsulosin hydrochloride (0.5 mg/0.2 mg). Each capsule will contain dutasteride (0.5 mg) (CJ) and tamsulosin pellets (0.2 mg) version 1.
Drug: Treatment sequence B — FDC 2 - Fixed dose combination capsule of dutasteride and tamsulosin hydrochloride (0.5 mg/0.2 mg). Each capsule will contain dutasteride (0.5 mg) (CL) and tamsulosin pellets (0.2 mg) version 2.
Drug: Treatment sequence C — Co-administration of dutasteride 0.5 mg capsule (Oblong, size 6, dull yellow capsules: Commercially available) and tamsulosin hydrochloride 0.2 mg tablet (White, round standard convex tablet: Commercially available).

SUMMARY:
This study will be an open-label, randomized, single dose, three way crossover study in healthy male subjects. The aim of the study is to evaluate the pharmacokinetic parameters of two formulations of a fixed dose combination (FDC) capsule of dutasteride and tamsulosin hydrochloride (HCl) (0.5 milligram [mg]/0.2 mg) relative to co-administration of dutasteride 0.5 mg capsules and tamsulosin hydrochloride 0.2 mg tablets in both the fed and fasted states. Approximately 84 healthy adult male subjects will be enrolled into the study and split into two cohorts (fed and fasted), allowing for approximately 36 subjects to complete each cohort. Subjects from both cohorts will receive single oral doses in 3 treatment periods and be randomized to one of six different treatment sequences (ABC, ACB, BAC, BCA, CAB, CBA) wherein A= FDC1: Dutasteride and tamsulosin HCl (0.5 mg/0.2 mg), B= FDC2: Dutasteride and tamsulosin HCl (0.5 mg/0.2 mg), C= Co-administration of commercial formulations of dutasteride(0.5mg) and tamsulosin HCl (0.2mg). Each treatment period will be separated by a minimum 28 day washout period. Blood samples for pharmacokinetic analysis will be taken at regular intervals after dosing. Safety will be assessed by measurement of blood pressure, heart rate and review of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Males aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator, in consultation with the GSK Medical Monitor if required, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilogram (kg) and body mass index (BMI) within the range 18 - 32 kg/m^2 (square meter) (inclusive).
* Male subjects with female partners of child-bearing potential must agree to use a condom. This criterion must be followed from the time of the first dose of study medication until 50 days post-last dose.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Able to swallow and retain oral medication.
* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) <2x (Upper limit of normal) ULN; alkaline phosphatase and bilirubin <=1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on single or averaged corrected QT (QTc) values of triplicate electrocardiograms (ECGs) obtained over a brief recording period: QT duration corrected for heart rate by Fridericia's formula (QTcF) <450 milliseconds (msec)

Exclusion Criteria:

Criteria Based Upon Medical Histories

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation.
* History of postural hypotension, dizziness, poor hydration, vertigo, vaso-vagal reactions or any other signs and symptoms of orthostasis, which in the opinion of the investigator could be exacerbated by tamsulosin and result in putting the subject at risk of injury.
* History of regular alcohol consumption within 6 months of the study defined for US sites as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 gram (g) of alcohol: 12 ounces (360 millilitre [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of diabetes or peptic ulcer disease which is uncontrolled by medical management.
* History of breast cancer or clinical breast examination finding suggestive of malignancy. History of malignancy within the past five years, except for basal cell carcinoma of the skin. Subjects with a prior malignancy who have had no evidence of disease for at least the past 5 years are eligible.
* Prior medical history or evidence of prostate cancer (e.g., positive biopsy, or suspicious ultrasound, or suspicious digital rectal examination [DRE]). Patients with suspicious ultrasound or DRE who have had a negative biopsy within the preceding 6 months and stable prostate specific antigen (PSA) are eligible for the study. Note: The investigator should make every appropriate effort to exclude the possibility of prostate cancer, including consideration of prostate biopsy in any subject with a known abnormal PSA.

Criteria Based Upon Diagnostic Assessments

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening;
* A positive pre-study drug/alcohol screen.
* A positive test for Human Immunodeficiency Virus (HIV) antibody. Other Criteria
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-07-10 (Actual); Primary Completion 2015-02-23 (Actual); Study Completion 2015-02-23 (Actual)

PRIMARY OUTCOMES:
Area under the curve from 0 to the time of the last quantifiable concentration (AUC[0-t]) of tamsulosin in serum | Pre-dose and post dose at 15 minutes (min), 30 min, 45 min, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours (h).
  Relative bioavailability of tamsulosin will be assessed by evaluating AUC (0-t).
Area under the curve from 0 to infinity (AUC[0-infinity]) of tamsulosin in serum | Pre-dose and post dose at 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 h post dose.
  Relative bioavailability of tamsulosin will be assessed by evaluating AUC (0-infinity).
Maximum drug concentration (Cmax) of dutasteride in serum | Pre-dose and post dose at 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 h post dose.
  Relative bioavailability of dutasteride will be assessed by evaluating Cmax
AUC(0-t) of dutasteride in serum | Pre-dose and post dose at 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 h post dose.
  Relative bioavailability of dutasteride will be assessed by evaluating AUC(0-t)

SECONDARY OUTCOMES:
Time to reach maximum serum concentration (tmax) of tamsulosin and dutasteride in serum | Pre-dose and post dose at 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 h post dose
  Pharmacokinetics of dutasteride and tamsulosin will be characterised by measuring tmax.
Terminal half-life (t½) of tamsulosin in serum (as data permit). | Pre-dose and post dose at 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 h post dose
  Pharmacokinetics of dutasteride and tamsulosin will be characterised by measuring t½
Safety and tolerability as assessed by Vital signs (blood pressure and pulse rate [PR]) | Up to Day 110
  Vital sign measurements will be measured in supine position after 5 minutes rest and will include systolic and diastolic blood pressure and pulse rate. Baseline for vital signs will be defined as the mean of the two blood pressure and pulse readings on Day -1.
Safety and tolerability as assessed by electrocardiogram (ECG) measurements | Up to Day 110
  Single 12-lead ECGs will be obtained at each time point during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT duration corrected for heart rate by Fridericia's formula (QTcF) intervals. Baseline for ECG will be defined as the mean of three measurements on Day -1
Safety and tolerability as assessed by review of adverse events (AEs) | Up to Day 110
  AEs will be collected from the start of dosing with Investigational Product and until the follow-up visit
Safety and tolerability as assessed by clinical laboratory safety data | Up to Day 56
  Clinical laboratory tests will include hematology, clinical chemistry and urinalysis

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Burns O, Zhu J, Manyak MJ, Ravindranath R, Koosha F, Haque N, Chung S. Relative Bioavailability of Fixed-Dose Combinations of Tamsulosin and Dutasteride: Results From 2 Randomized Trials in Healthy Male Volunteers. Clin Pharmacol Drug Dev. 2018 May;7(4):422-434. doi: 10.1002/cpdd.380. Epub 2017 Aug 11. PMID 28800206
- See also: Results for study 117057 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/117057?search=study&search_terms=117057#rs
- Available data/document: Annotated Case Report Form: 117057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 117057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 117057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 117057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 117057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 117057 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register